CLINICAL TRIAL: NCT01864577
Title: Efficacy of Negative Pleural Suction in Tube Thoracostomy for Patients With Penetrating and/or Blunt Chest Trauma: a Randomized Clinical Trial
Brief Title: Negative Pleural Suction for Tube Thoracostomy in Patients With Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Hospital San Vicente Fundación (Other)
Responsible Party: Principal Investigator, Camila Mejia, Surgical Resident, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01UDEACx2013
Record Dates: First submitted 2013-05-20; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Hemothorax; Pneumothorax; Hemopneumothorax; Chest Injury Trauma Blunt; Chest Injury Trauma; Chest Injury Penetrating Wound
MeSH Terms: conditions — Hemothorax; Pneumothorax; Hemopneumothorax

ARMS (2):
- With negative pleural suction (Experimental): Patients are put on negative pleural suction at - 20 cm H2O
  Interventions: Other: Negative Pleural Suction at -20 cm H2O; Other: Water seal
- With water seal (Active Comparator): Patients al left on water seal only
  Interventions: Other: Water seal

INTERVENTIONS:
Other: Negative Pleural Suction at -20 cm H2O
  Arms: With negative pleural suction
Other: Water seal

SUMMARY:
The purpose of this study is to determine whether the use of negative pleural suction in tube thoracostomy is more effective than water seal alone for the treatment of pneumothorax and/or hemothorax in patients with chest trauma.

ELIGIBILITY:
Inclusion Criteria:

* Pneumothorax after penetrating o blunt chest trauma
* Hemothorax after penetrating o blunt chest trauma
* Hemopneumothorax after penetrating o blunt chest trauma
* Require tube thoracostomy

Exclusion Criteria:

* Invasive mechanical ventilation
* Emergent Surgery (thoracoscopy, open thoracotomy)
* Chronic pulmonary diseases (COPD, CRPD)
* Severe traumatic brain injury
* Glasgow coma scale upon arrival <8/15

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Lenght of Hospital stay | 30 days

SECONDARY OUTCOMES:
Incidence of persistent bronchopleural fistulae | 30 days
Incidence of coagulated Hemothorax | 30 days
Incidence of empyema | 30 days
Incidence of recurrent pneumothorax | 30 days
Number of patients necessitating surgical interventions (includes new thoracostomy, thoracoscopy and open thoracotomy) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Camila Mejia, Resident, General Surgery, Principal Investigator — Universidad de Antioquia
Locations (1):
- Departamento de Cirugía, Universidad de Antioquia, San Vicente Fundación Hospital Universitario, Medellín, Antioquia, Colombia